CLINICAL TRIAL: NCT01601548
Title: Cancer and Mindfulness-Based Cancer Recovery After Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2012NTLS014
Record Dates: First submitted 2012-04-24; First posted 2012-05-18 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Breast Cancer; Colorectal Cancer; Ovarian Cancer; Uterine Cancer
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Ovarian Neoplasms; Uterine Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Arm (Experimental): Subjects are randomized to the Mindfulness Based Cancer Recovery (MBSR) intervention. Participants are presented with mindfulness medication techniques and share their experiences related to these meditation practices. There is a home practice component with an expectation of regular home meditation practice of 45 minutes per day. A full day silent retreat will occur in the second half of the course, providing an opportunity for class participants to gain experience with mindfulness techniques.
  Interventions: Behavioral: Mindfulness Based Cancer Recovery
- Control Arm (No Intervention): No intervention is administered. Health-related quality of life questionnaires will be completed.

INTERVENTIONS:
Behavioral: Mindfulness Based Cancer Recovery — Defined as practices or interventions that focus on the connection and integration of the mind and body and the ability for these connections to effect changes on physical, emotional and spiritual levels for the purpose of promoting health and well being. MBCR is a psycho-educational program developed by Dr. Linda Carlson. It is a step by step mindful-based stress reduction program (MBSR) designed to help cancer patients cope with their cancer diagnosis and treatment
  Arms: Intervention Arm

SUMMARY:
Upon the completion of aggressive chemotherapy and radiation for curative intent cancers, many cancer survivors suffer from a myriad of symptoms ranging from physical symptoms such as hot flashes, insomnia, and fatigue to psychosocial symptoms including depression and anxiety. Mindfulness Based Cancer Recovery (MBCR) is a type of mind-body intervention. Mind-body interventions are defined as practices or interventions that focus on the connection and integration of the mind and body and the ability for these connections to effect changes on physical, emotional and spiritual levels for the purpose of promoting health and well being.

DETAILED DESCRIPTION:
MBCR is a step wise standardized behavioral intervention of MBSR. The program is usually conducted in eight weekly class sessions that are 2-2.5 hours in length. During class sessions, participants are presented with mindfulness meditation techniques and share their experiences related to these meditation practices. There is a home practice component with an expectation of regular home meditation practice of 45 minutes per day. In addition to home meditation practice there are often reading assignments and reflective exercises that relate to mindfulness. A full day retreat generally occurs in the second half of the course, providing an opportunity for class participants to gain extended experience with mindfulness techniques.

ELIGIBILITY:
Inclusion Criteria:

* Stage I-III breast cancer, gynecologic cancer or colorectal cancer
* Cancer survivor at least 18 years of age at the time of study enrollment
* Completed chemotherapy within the past six months at the time of consent (adjuvant hormone therapy is allowed)

Exclusion Criteria:

* Psychologic disease in which informed consent cannot be obtained from the subject
* Need for ongoing chemotherapy and/or radiation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2012-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Change in Medical Outcomes Study Scores - Intervention versus Control | Day 1, Week 8 and 4 Month Follow-Up
  MOS SF-36: Medical Outcomes Study 36-Item Short-Form

SECONDARY OUTCOMES:
Change in Functional Assessment in Cancer Therapy Fatigue Scores - Intervention versus Control | Day 1, Week 8 and 4 Month Follow-Up
  FACT-F: Functional Assessment in Cancer Therapy - Fatigue
Change in Pittsburgh Sleep Quality Index Scores - Intervention versus Control | Day 1, Week 8 and 4 Month Follow-Up
  PSQI: Pittsburgh Sleep Quality Index
Change in State-Trait Anxiety Inventory Scores - Intervention versus Control | Day 1, Week 8 and 4 Month Follow-Up
  20-item State-Trait Anxiety Inventory
Comparison of Sexual Functioning Scale Scores - Intervention versus Control | Day 1, Week 8 and 4 Month Follow-Up
  MOS Sexual Functioning Scale
Change in Self-Compassion Scale Scores - Intervention versus Control | Day 1, Week 8 and 4 Month Follow-Up
  SCS-SF: Self-Compassion Scale - Short Form
Change in Self-Collected Information - Intervention versus Control | Day 1, Week 8 and 4 Month Follow-Up
  Self collected and self-report information regarding weekly meditation practice time, recorded class attendance and information from participants regarding barriers and challenges to practice, and perceived benefits to practice will be collected.
Change in Number of Natural Killer Cells - Intervention versus Control | Day 1, Week 8 and 4 Month Follow-Up

CONTACTS AND LOCATIONS:
Overall Officials: Anne Blaes, M.D., Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States